CLINICAL TRIAL: NCT04844710
Title: The Effects of Combined Treatment of Acupuncture Intervention & Standard of Care on Laboratory and Clinical Outcomes in Hospitalized COVID-19 Patients With Mild-Moderate Symptoms
Brief Title: The Effects of Acupuncture in Overcoming Inflammatory Response to COVID-19 Mild-moderate Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, dr. Dwi Rachma Helianthi, Sp.Ak, Principal Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KET-845/UN2.F1/ ETIK/PPM.2020
Record Dates: First submitted 2021-04-12; First posted 2021-04-14 (Actual); Last update posted 2021-04-14 (Actual); Status verified 2021-04

CONDITIONS: Acupuncture; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Acupuncture Therapy; Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Manual acupuncture and standard care
  Interventions: Combination Product: acupuncture and standard care
- Control (Other): Standard care only
  Interventions: Drug: standard care

INTERVENTIONS:
Combination Product: acupuncture and standard care — manual acupuncture in acupoint LI4, LI11, ST36 every 2 days for 6 times standard care
  Other Names: Combined Treatment of Acupuncture Intervention and Standard of Care
  Arms: Treatment
Drug: standard care — standard care only
  Other Names: standard of care COVID-19
  Arms: Control

SUMMARY:
Coronavirus disease 2019 (COVID-19) is a problem that is being faced in more than 200 countries in the world, including Indonesia. The World Health Organization (WHO) has declared the COVID-19 outbreak as a pandemic. The transmission of the virus occurred rapidly that 2 weeks from the first case diagnosed, 1000 patients tested positive. A week later, the number of positive cases exceeded 4600, reaching more than 30,000 patients and 2,500 deaths on March 18, 2020. The death rate due to COVID-19 in Indonesia is one of the highest in Asia.

To date, no therapy has been shown to be effective for Coronavirus (SARS-CoV-2). A vaccine for SARS-CoV-2 also has not been found at this time and is in the research phase. Current management of COVID-19 patients focuses primarily on providing supportive care. Currently, several countries make treatment guidelines for COVID-19 patients by providing several types of anti-viral drugs and other drugs such as chloroquine or hydroxychloroquine, immunoglobulins, anti-cytokine agents or immunomodulators.

The administration of these drugs does not escape the various side effects experienced by patients. Administration of chloroquine or hydroxychloroquine carries the risk of causing prolonged QT interval which can lead to arrhytmia disturbances such as torsades des pointes in certain people. Administration of chloroquine or hydroxychloroquine in combination with azithromycin increases the risk of developing arrhythmias. Giving anti-viruses such as lopinavir / ritonavir, umifenovir, remdesivir, favipiravir can also cause various side effects including gastrointestinal disturbances (nausea, vomiting, diarrhea), impaired liver function, and hyperuricaemia. Treatment with human immunoglobulins has been associated with a significantly increased risk of thrombotic events.

Currently, no acupuncture research on COVID-19 patients has been published. However, acupuncture can play a role in several conditions that occur in COVID-19 according to the pathophysiology that occurs, this has been proven through several clinical studies conducted on non-COVID-19 cases that have pathophysiology that resemble COVID-19 conditions. In COVID-19 with mild-moderate symptoms, acupuncture can play a role in boosting the immune system, including increasing the number of Natural Killer cells and lymphocytes. Whereas in cases of severe COVID-19 symptoms, it is hoped that acupuncture can provide anti-inflammatory effect and prevent cytokine storm.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 18 years of age, COVID-19 confirmed by RT-PCR with mild-moderate symptoms
* Willing to participate in research.
* Willing to follow the research process to completion.

Exclusion Criteria:

* The patient has contraindications to acupuncture (medical emergencies, pregnancy, malignancy, blood clotting disorders and consumption of anti-coagulant drugs).
* Patients with myeloproliferative disorders.
* There is a tumor or infection in the area where the acupuncture point is inserted.
* Patients with a history of uncontrolled Diabetes Mellitus with random blood sugar levels > 200 mg / dL

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Changes of percentage of lymphocyte count | before treatment and after 2 weeks of treatment
  Changes of percentage of lymphocyte count (diff count) between before treatment and after 2 weeks of treatment (after sixth acupuncture session given)
Changes of Erythrocyte sedimentation rate | before treatment and after 2 weeks of treatment
  Changes of Erythrocyte sedimentation rate between before treatment and after 2 weeks of treatment (after sixth acupuncture session given)
Changes of Ferritin level | before treatment and after 2 weeks of treatment
  Changes of Ferritin level between before treatment and after 2 weeks of treatment (after sixth acupuncture session given)
Changes of C-Reactive Protein level | before treatment and after 2 weeks of treatment
  Changes of C-reactive protein level between before treatment and after 2 weeks of treatment (after sixth acupuncture session given)
Clinical changes | before treatment and after 2 weeks of treatment
  duration of cough and fever during the patients are hospitalized

CONTACTS AND LOCATIONS:
Overall Officials: Dwi Rachma Helianthi, MD, Principal Investigator — Indonesia University
Locations (1):
- Medical Acupuncture Department FKUI-RSCM, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No